CLINICAL TRIAL: NCT05370521
Title: A Randomized, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety and Efficacy of Tildacerfont in Adult Subjects With Polycystic Ovary Syndrome (PCOS) and Elevated Adrenal Androgens
Brief Title: A Study of Safety and Efficacy of Tildacerfont in Females With Polycystic Ovary Syndrome and Elevated Adrenal Androgens
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was discontinued early by the sponsor
Sponsor: Spruce Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPR001-210
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; Elevated Adrenal Androgen; Adrenal Disorder; Polycystic Ovary Syndrome; Womens health
MeSH Terms: conditions — Polycystic Ovary Syndrome; Adrenal Gland Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind randomization performed by IRT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment with Tildacerfont (Experimental): Subjects randomized in this arm received 4 weeks of 50 mg of oral tildacerfont tablet, followed by 4 weeks of 100 mg oral tildacerfont tablet, and then 4 weeks of 200 mg oral tildacerfont tablet for a total of 12 weeks of treatment.
  Interventions: Drug: Tildacerfont
- Placebo Control Arm (Placebo Comparator): Subjects randomized in this arm received 12 weeks of oral matched-placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tildacerfont — Oral tablet formulation taken once daily.
  Other Names: SPR001
  Arms: Treatment with Tildacerfont
Drug: Placebo — Non-active dosage form taken once daily.
  Arms: Placebo Control Arm

SUMMARY:
An investigation of the safety and efficacy of tildacerfont in women with PCOS and elevated adrenal androgens

DETAILED DESCRIPTION:
This was a phase 2 study to evaluate the efficacy, safety and tolerability of 3 doses of tildacerfont in approximately 39 women with PCOS and elevated adrenal androgens assessed by elevated DHEAS levels. Subjects were randomized 2:1 (tildacerfont:placebo) at baseline. The study consisted of 3 consecutive 4-week treatment periods at each dose level. Duration of participation was approximately 25 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 18 to 40 years old at Screening visit
* Diagnosis of PCOS (either historical or during Screening) according to NIH (1990) criteria
* DHEAS level > age-matched upper limit of normal (ULN) at Screening visit
* Agree to follow industry standard contraception guidelines within protocol

Exclusion Criteria:

* Evidence of:

  1. History of congenital adrenal hyperplasia (CAH), Cushing's syndrome, pituitary or adrenal disease
  2. Clinically significant hyperprolactinemia
  3. Thyroid stimulating hormone (TSH) <0.1 mU/mL or >4.5mU/mL at Screening
  4. Cortisol levels concerning for adrenal insufficiency
  5. Other findings suggestive of secondary cause for anovulation and/or hyperandrogenemia
* Total testosterone levels >140 ng/dL, DHEAS >650 mcg/dL, virilization or other signs or symptoms concerning for ovarian hyperthecosis or androgen-secreting tumors
* Medical conditions that require glucocorticoid treatment within 30 days of screening and throughout the duration of the study
* Clinically significant unstable medical conditions, illness, or chronic diseases
* Prior hysterectomy or bilateral oophorectomy
* Females who are pregnant or nursing

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility for females is based on gender assignment at birth.
Enrollment: 27 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Will Charlton, MD, Study Director — Spruce Biosciences
Locations (20):
- United States (20):
  - Spruce Study Site, Sacramento, California
  - Spruce Study Site, San Francisco, California
  - Spruce Study Site, New Haven, Connecticut
  - Spruce Study Site, Clearwater, Florida
  - Spruce Study Site, Lake Worth, Florida
  - Spruce Study Site, Miami, Florida
  - Spruce Study Site, Winter Park, Florida
  - Spruce Study Site, Idaho Falls, Idaho
  - Spruce Study Site, Wichita, Kansas
  - Spruce Study Site, Boston, Massachusetts
  - Spruce Study Site, Fall River, Massachusetts
  - Spruce Study Site, Southfield, Michigan
  - Spruce Study Site, Williamsville, New York
  - Spruce Study Site, Raleigh, North Carolina
  - Spruce Study Site, Cincinnati, Ohio
  - Spruce Study Site, Cleveland, Ohio
  - Spruce Study Site, Philadelphia, Pennsylvania
  - Spruce Study Site, Bedford, Texas
  - Spruce Study Site, Houston, Texas
  - Spruce Study Site, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 82 subjects that were screened, a total of 27 subjects enrolled in the study (10 subjects in the placebo arm and 17 subjects in the tildacerfont arm).
Groups:
- Treatment With Tildacerfont: Subjects randomized in this arm received 4 weeks of 50mg of oral tildacerfont tablet, followed by 4 weeks of 100 mg oral tildacerfont tablet, and then 4 weeks of 200 mg oral tildacerfont tablet for a total of 12 weeks of treatment.
Period: Overall Study
Arm/Group | Treatment With Tildacerfont | Placebo Control Arm
Started | 17 | 10
Completed | 16 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment With Tildacerfont: Subjects randomized in this arm will receive 4 weeks of 50mg of oral tildacerfont tablet, followed by 4 weeks of 100 mg oral tildacerfont tablet, and then 4 weeks of 200 mg oral tildacerfont tablet for a total of 12 weeks of treatment.
- Placebo Control Arm: Subjects randomized in this arm will receive 12 weeks of oral matched-placebo tablet
- Total: Total of all reporting groups
Arm/Group | Treatment With Tildacerfont | Placebo Control Arm | Total
Number analyzed (Participants) | 17 | 10 | 27
Age, Categorical [Count of Participants; unit: Participants] — Female subjects aged 18 to 40 years old due to the nature of the disease
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 17 | 10 | 27
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 27
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 15 | 9 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 10 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0
Dehydroepiandrosterone sulfate (DHEAS) [Mean (Standard Deviation); unit: ug/dL] | 351.3 (90.53) | 387.8 (107.16) | 364.8 (96.65)
Adrenocorticotropic hormone (ACTH) [Mean (Standard Deviation); unit: pg/dL] | 23.88 (11.927) | 22.3 (12.013) | 23.27 (11.744)
17-hydroxyprogesterone (17-OHP) [Mean (Standard Deviation); unit: ng/dL] | 83.2 (86.28) | 62.1 (54.1) | 75.4 (75.51)
Androstenedione (A4) [Mean (Standard Deviation); unit: ng/dL] | 185.2 (75.19) | 130.0 (65.96) | 166.8 (75.61)
Testosterone [Mean (Standard Deviation); unit: ng/dL] | 61.0 (21.97) | 61.1 (26.97) | 61.0 (23.43)
Cortisol [Mean (Standard Deviation); unit: ug/dL] | 13.44 (4.847) | 16.41 (7.206) | 14.54 (5.879)

OUTCOME MEASURES:

1. Secondary Outcome: Reduction in DHEAS
Description: Number of subjects with >/=30% change from baseline in DHEAS
Time Frame: 12 weeks (assessed at Baseline, Weeks 4, 8 and 12)
Population: Number of subjects with a >/=30% change from Baseline in DHEAS (μg/dL) at Week 12, Modified Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment With Tildacerfont: Subjects randomized in this arm will receive 4 weeks of 50 mg of oral tildacerfont tablet, followed by 4 weeks of 100 mg oral tildacerfont tablet, and then 4 weeks of 200 mg oral tildacerfont tablet for a total of 12 weeks of treatment.
Arm/Group | Treatment With Tildacerfont | Placebo Control Arm
Number analyzed (Participants) | 16 | 10
Participants | 1 | 1

2. Secondary Outcome: Normalization of DHEAS
Description: Number of subjects with DHEAS =/< upper limit of normal for DHEAS
Time Frame: 12 weeks (assessed at Baseline, Weeks 4, 8 and 12)
Population: Number of subjects with DHEAS =/< upper limit of normal for DHEAS at Week 12, Modified Intent-to-treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Tildacerfont | Placebo Control Arm
Number analyzed (Participants) | 16 | 10
Participants | 8 | 6

3. Secondary Outcome: Number of Subjects With TEAE as Assessed by CTCAE Version 5
Description: Evaluation of safety of tildacerfont with PCOS as measured by number of subjects with adverse events following dosing by CTCAE Version 5
Time Frame: 12 weeks (assessed at Baseline, Weeks 4, 8 and 12)
Population: All subjects who received at least 1 dose of placebo or tildacerfont; Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Tildacerfont | Placebo Control Arm
Number analyzed (Participants) | 17 | 10
Participants | 13 | 9

4. Primary Outcome: Change in DHEAS
Description: To evaluate the effect of tildacerfont in changing (reducing) DHEAS in subjects with PCOS and elevated adrenal androgens
Time Frame: 12 weeks (assessed at Baseline, Weeks 4, 8 and 12)
Population: Analysis of Change from Baseline in DHEAS (μg/dL) at Week 12, Modified Intent-to-Treat Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/dL
Groups:
- Treatment With Tildacerfont: Subjects randomized in this arm rfeceived 4 weeks of 50 mg of oral tildacerfont tablet, followed by 4 weeks of 100 mg oral tildacerfont tablet, and then 4 weeks of 200 mg oral tildacerfont tablet for a total of 12 weeks of treatment.
Arm/Group | Treatment With Tildacerfont | Placebo Control Arm
Number analyzed (Participants) | 16 | 10
ug/dL | -22.93 (67.600) | -7.56 (16.00)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events are presented as totals for subjects receiving tildacerfont and are not separated by dose level.
Arm/Group | Treatment With Tildacerfont | Placebo Control Arm
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/10
Other Adverse Events (participants affected / at risk) | 13/17 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Tildacerfont (N=17) | Placebo Control Arm (N=10)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Tildacerfont (N=17) | Placebo Control Arm (N=10)
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 8 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
COVID-19 (Infections and infestations) | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Viral rhinitis (Infections and infestations) | 1 | 0
Blood potassium increased (Investigations) | 0 | 1
Total bile acids increased (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Tension headache (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Pruitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor; therefore, there were a small number of subjects for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT05370521/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT05370521/SAP_001.pdf
  • Informed Consent Form (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT05370521/ICF_002.pdf